CLINICAL TRIAL: NCT07099599
Title: Image Detection of Impaired Microcirculatory Reperfusion
Acronym: ID IMR
Status: Recruiting | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Yasmin Aziz, Principal Investigator, University of Cincinnati
Other Study IDs: 2024-0526; 24CDA1268532 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2025-03-16; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Ischemic Stroke, Acute; Large Vessel Occlusion
Keywords: No Reflow; Microcirculatory Reperfusion; Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Thrombectomy-Treated Subjects with Anterior Circulation Vessel Occlusion: Patients with anterior circulation LVO or equivalent stroke treated with mechanical thrombectomy.
  Interventions: Diagnostic Test: CT Perfusion

INTERVENTIONS:
Diagnostic Test: CT Perfusion — CT perfusion within 90 minutes of complete angiographic reperfusion

SUMMARY:
Stroke affects one patient every 40 seconds in the United States. It is most commonly caused by blood clots that develop in the blood vessels of the brain. These blood clots interrupt the normal flow of blood and oxygen to the nerve cells in the brain. When this occurs, the nerve cells can die, causing permanent damage to that area of the brain. That damage can result in loss of normal function to a patient's vision, strength, sensation, balance, or speech. These changes can remain permanent if blood flow is not restored to the brain. Thankfully, there are treatments available to help get rid of these blood clots. One of these treatments is a procedure to physically remove the blood clot causing stroke. This practice is now routinely done at all major stroke centers.

Special imaging for stroke is now available at these major stroke centers. This imaging looks at blood flow in and around the area of brain that is dying. By performing these scans after the procedure, we can see that not all of brain is being saved by the procedure. That is a problem, because we know that saving brain cells can make a big difference in how patients recover from stroke. The purpose of this study is to determine which brain tissue will not get saved by blood clot removal. We will do this by using specialized imaging after the procedure. The study will discover if there is more brain tissue that can be saved after the procedure. Once we can determine this, our next steps will be looking at ways to save this tissue in the studies that follow. For example, we will look to see if medications can be given after the procedure to help save those brain areas. This study lays the groundwork for future studies to help save all the brain tissue we possibly can from dying during the stroke. This is our best chance of getting all patients affected by stroke the opportunity to live their best lives after stroke.

DETAILED DESCRIPTION:
Image Detection of Impaired Microcirculatory Reperfusion (ID IMR) is a single center, prospective, feasibility study. It is designed to test the feasibility of utilizing post-thrombectomy CT Perfusion to identify a radiographic biomarker of IMR as well as other key variables associated with infarct expansion following complete angiographic reperfusion from thrombectomy in large vessel occlusion (LVO) stroke. The best biomarker identified from this study will be validated in a larger prospective study as a surrogate biomarker of IMR in LVO stroke.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than or equal to 18 years of age
* Last known normal (LKN) within 24 hours
* Ischemic stroke due to anterior circulation LVO (intracranial internal carotid artery [ICA], proximal middle cerebral artery [M1], M1/M2 bifurcation, or proximal dominant M2 occlusion)
* mTICI2c or mTICI3 on digital subtracted angiography (DSA) following mechanical thrombectomy

Exclusion Criteria:

* Significant renal insufficiency (glomerular filtration rate <30mg/ml/min2 while not on dialysis)
* Contraindication to iodinated contrast
* Contraindication to magnetic resonance imaging (e.g., pacemaker incompatibility)
* Prior significant stroke in same vascular territory ipsilateral stroke
* Tandem vessel occlusion (i.e., extracranial ICA and ipsilateral intracranial M1/M2 occlusion)
* Greater than 4 clot retrieval attempts
* Enrollment in another acute stroke interventional study (with the exception of thrombectomy device registries)
* Pregnancy
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thrombectomy-treated subjects with mTICI2c or 3 reperfusion of a previously occluded anerior circulation vessel.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of 90-minute CTP and 48-96-hr MRI | From enrollment to 96 hours
  The primary outcome is feasibility determined by greater than or equal to 80% of the planned sample size for whom technically adequate 90-minute CTP and 48-96 hour MRI key parameters (baseline penumbra volume [Tmax greater than 4 seconds], predicted infarct core volume [CBF greater than 30%], and follow-up infarct volume [MRI DWI]) are usable.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Perfusion parameters from CTP
Time Frame: All data will be available in an AHA-approved repository 1 year after conclusion of funding period
Access Criteria: Data will be shared upon reasonable request